CLINICAL TRIAL: NCT05113550
Title: Surgical Treatment of Hepatic Hydatidosis in Elderly Patients
Acronym: ELDHIDA
Status: Completed | Type: Observational
Sponsor: Universidad de Extremadura (Other)
Responsible Party: Principal Investigator, Gerardo Blanco-Fernández, Profesor, Universidad de Extremadura
Other Study IDs: HUB-2021-01
Record Dates: First submitted 2021-10-28; First posted 2021-11-09 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-10

CONDITIONS: Cystic Echinococcosis
MeSH Terms: conditions — Echinococcosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Young group: patients < 70 years of age
  Interventions: Other: Surgical remove
- Elderly: Patients ≥ 70 years of age)
  Interventions: Other: Surgical remove

INTERVENTIONS:
Other: Surgical remove — liver hydatid cyst (LHC) treated by total or partial pericystectomy

SUMMARY:
Cystic echinococcosis is a clinically complex chronic parasitic disease and a major socioeconomic problem in endemic areas. The safety of liver resection in elderly patients is often debated among medical professionals. The investigators analyzed the postoperative morbidity and mortality rates of elderly patients who underwent surgery at our unit.

DETAILED DESCRIPTION:
Retrospective observational study from prospective database focused on liver hydatidosis carried out at our Hepato-Pancreato-Biliary Surgery Unit. The study period spanned from January 2006 to October 2020. The study was approved by the Research Ethics Committee of our hospital. An informed consent from the patient was not required since the study was retrospective and observational, and entailed no risk. Seventy years of age was the cutoff age to consider patients as elderly.

Inclusion criteria of patients: liver hydatid cyst (LHC) diagnosed by preoperative computed tomography (CT) or magnetic resonance imaging (MRI) and pathological diagnosis after surgery, and LHC treated by total or partial pericystectomy.

Exclusion criteria of patients: emergency surgery and simple drainage of cyst.

ELIGIBILITY:
Inclusion Criteria:

* liver hydatid cyst (LHC)
* pathological diagnosis after surgery
* LHC treated by total or partial pericystectomy

Exclusion Criteria:

* emergency surgery and simple drainage of cyst

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with liver hydatidosis carried out at our Hepato-Pancreato-Biliary Surgery Unit
Sampling Method: Non-Probability Sample
Enrollment: 279 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Morbidity | 90 days
  Patients with postoperative morbidity according to the Clavien-Dindo score 19, "severe complication" (Clavien-Dindo ≥ IIIa) and postoperative mortality

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo Blanco-Fernández, MD, PhD, Principal Investigator — University of Extremadura
Locations (2):
- Spain (2):
  - Universidad de Extremadura- Facultad de Medicina, Badajoz
  - Gerardo Blanco-Fernández, Badajoz

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mihmanli M, Idiz UO, Kaya C, Demir U, Bostanci O, Omeroglu S, Bozkurt E. Current status of diagnosis and treatment of hepatic echinococcosis. World J Hepatol. 2016 Oct 8;8(28):1169-1181. doi: 10.4254/wjh.v8.i28.1169. PMID 27729953
- [Background] Adamina M, Guller U, Weber WP, Oertli D. Propensity scores and the surgeon. Br J Surg. 2006 Apr;93(4):389-94. doi: 10.1002/bjs.5265. PMID 16400708
- [Background] Jaen-Torrejimeno I, Lopez-Guerra D, Prada-Villaverde A, Blanco-Fernandez G. Pattern of Relapse in Hepatic Hydatidosis: Analysis of 238 Cases in a Single Hospital. J Gastrointest Surg. 2020 Feb;24(2):361-367. doi: 10.1007/s11605-019-04163-7. Epub 2019 Feb 26. PMID 30809783
- [Background] Jaen-Torrejimeno I, Latorre-Fragua R, Lopez-Guerra D, Rojas-Holguin A, Manuel-Vazquez A, Blanco-Fernandez G, Ramia JM. Jaundice as a clinical presentation in liver hydatidosis increases the risk of postoperative biliary fistula. Langenbecks Arch Surg. 2021 Jun;406(4):1139-1147. doi: 10.1007/s00423-020-02070-z. Epub 2021 Jan 2. PMID 33389115
- [Result] Muhtarov M, Rainova I, Tamarozzi F. Treatment of Hepatic Cystic Echinococcosis in Patients from the Southeastern Rhodope Region of Bulgaria in 2004-2013: Comparison of Current Practices with Expert Recommendations. Am J Trop Med Hyg. 2016 Apr;94(4):900-5. doi: 10.4269/ajtmh.15-0620. Epub 2016 Feb 1. PMID 26834196